CLINICAL TRIAL: NCT00097487
Title: Clinical Outcomes in Patients With HER2 Gene-Amplified Metastatic Breast Cancer Treated With First Line Herceptin in Combination With a Taxane: A Phase IV, Prospective, Community Based Study
Brief Title: A Study of Patients With HER2 Gene Amplified Metastatic Breast Cancer Treated With First Line Herceptin and a Taxane
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Other Study IDs: H2251n
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer; Metastases
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study is a Phase IV, prospective, nonrandomized, community-based study of clinical outcomes in patients with metastatic breast cancer treated with Herceptin and a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Available tissue for central laboratory evaluation of HER2 status
* Histologically confirmed, measurable or nonmeasurable but evaluable, HER2 positive metastatic breast cancer (HER2 positive is defined as 3+ staining by IHC or gene amplification by FISH, determined by the local or central laboratory)
* Life expectancy >6 months
* Female, age >=18 years
* ECOG performance status of 0, 1, or 2
* Adequate bone marrow function as indicated by the following: *ANC >1500/uL, *Platelet count >=100,000/uL
* Adequate renal function, as indicated by creatinine <=1.5× upper limit of normal (ULN)
* Adequate liver function, as indicated by bilirubin <=1.5× ULN and AST or ALT <2× ULN unless related to primary disease
* Use of an adequate means of birth control (women of childbearing potential)

Exclusion Criteria:

* Initiation of Herceptin >=4 weeks after beginning taxane chemotherapy
* Prior chemotherapy for metastatic disease
* Prior cumulative anthracycline dose of >360 mg/m2
* History of significant cardiac disease or uncontrolled arrhythmias
* Ejection fraction of <50% or below the lower limit of normal
* Active infection
* Symptomatic or untreated brain metastases
* Pregnancy or lactation
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest
* Hypersensitivity to study medications
* Major organ failure or systemic disease precluding the safe administration of study medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2000-11-30 (Actual); Study Completion 2004-09-30 (Actual)